CLINICAL TRIAL: NCT00367094
Title: Efficacy and Safety of the Combination of Benazepril Plus Hydrochlorothiazide in Chinese Patients With Mild to Moderate Essential Hypertension Not Adequately Controlled With Benazepril
Brief Title: Combination of Benazepril Plus Hydrochlorothiazide in Chinese Patients With Mild to Moderate Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLHT344ACN01
Record Dates: First submitted 2006-08-21; First posted 2006-08-22 (Estimated); Last update posted 2007-07-09 (Estimated); Status verified 2007-03

CONDITIONS: Hypertension
Keywords: Hypertension, benazepril, hydrochlorothiazide, fixed combination
MeSH Terms: conditions — Hypertension | interventions — benazepril; Hydrochlorothiazide

INTERVENTIONS:
Drug: Benazepril plus hydrochlorothiazide

SUMMARY:
This study will evaluate efficacy and safety data for benazepril/hydrochlorothiazide in adult Chinese patients with mild to moderate essential hypertension. Patients whose blood pressure is not adequately controlled with benazepril monotherapy during a 4 week run-in period will be randomly allocated to double blind treatment over 8 weeks with either a combination of benazepril/hydrochlorothiazide per day or continuation of benazepril per day.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, age 18 or older
* Given informed consent
* Diagnosed as having mild to moderate essential hypertension

Exclusion Criteria:

* Severe hypertension
* Significant preexisting cardiovascular and cerebrovascular disease
* Diabetes mellitus type 1 or poorly controlled diabetes mellitus type II
* Advanced renal impairment

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296
Dates: Start 2006-07

PRIMARY OUTCOMES:
Change in diastolic blood pressure from baseline to week 8

SECONDARY OUTCOMES:
Change in systolic blood pressure from baseline to week 8
Proportion of patients with blood pressure less than 140/90 mmHg at week 8
Ambulant blood pressure monitoring profiles at baseline and week 8

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Principal Investigator — Novartis Pharmaceuticals
Locations (1):
- Novartis, Beijing, China